CLINICAL TRIAL: NCT04001153
Title: Occlusal Compensation After the Placement of Preformed Metal Crowns Using the Hall Technique for Carious Primary Molars; Where it Occurs and Clinical Implications
Brief Title: Occlusal Compensation After the Hall Technique
Acronym: CHAT
Status: Withdrawn | Type: Observational
Why Stopped: There will be no opportunity to recruit patients during the pandemic of COVID-19 and possibly even post-pandemic
Sponsor: University of Dundee (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nicola Innes, Professor of Paediatric Dentistry & Associate Dean for Teaching and Learning, University of Dundee
Other Study IDs: 1-006-19
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries
Keywords: Hall Technique; Primary Molar; Vertical Dimension
MeSH Terms: conditions — Dental Caries | interventions — Dental Impression Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Upper primary first molar: Children already treatment planned to have a Hall Technique crown placed to manage primary molars carious lesions will have dental impressions taken before the crown placement, immediately after and at 2, 4, 6 and 8 weeks follow-up.
  Interventions: Other: Dental impressions
- Lower primary first molar: Children already treatment planned to have a Hall Technique crown placed to manage primary molars carious lesions will have dental impressions taken before the crown placement, immediately after and at 2, 4, 6 and 8 weeks follow-up.
  Interventions: Other: Dental impressions
- Upper primary second molar: Children already treatment planned to have a Hall Technique crown placed to manage primary molars carious lesions will have dental impressions taken before the crown placement, immediately after and at 2, 4, 6 and 8 weeks follow-up.
  Interventions: Other: Dental impressions
- Lower primary second molar: Children already treatment planned to have a Hall Technique crown placed to manage primary molars carious lesions will have dental impressions taken before the crown placement, immediately after and at 2, 4, 6 and 8 weeks follow-up.
  Interventions: Other: Dental impressions

INTERVENTIONS:
Other: Dental impressions — Children will be included in this study if they already are treatment planned to receive a Hall Technique preformed metal crown (HTPMC) to manage carious lesions in primary molars. They will have a dental impression taken before and after the HTPMC placement to find out what happens with their bite after the treatment.
  The dental impressions will be cast up into stone study models so that we can track the changes that happens in children's bites after placing the HTPMC (as it increases the height of children's bite when placed) and let them know what to expect after this procedure and as part of this study, additional follow-ups will be required 2, 4, 6 and 8 weeks after the HTPMC placement to allow us to track the changes in the bite at regular intervals to see when the child's bite returns to its pre-treatment state.

SUMMARY:
The Hall Technique preformed metal crown (HTPMC) is used to treat decayed primary molars. The correct size is chosen and pushed over the tooth with no tissue removal. A side-effect of the HTPMC is the increasing of tooth's height changing the child's bite vertically, resulting in a premature contact on the crowned tooth. Clinical trials have looked at it and measured the initial and final vertical change (after the HTPMC placement) and have found that vertical dimension (VD) is re-established within a few weeks. They suggest that there might be a compensatory mechanism related to the crowned tooth/its opposing tooth. None of these trials measured how long it took the occlusion to return to its pre-crown state, merely observing at convenient follow-up times that it happens. Neither has there been any investigation into the mechanisms by which the compensation occurs.

A pilot trial was conducted at Dundee Dental School (DDS) in 2013 to find the best and most reproducible method to measure the change in VD after HTPMC placement. It compared 4 different approaches: direct clinical measurement; clinical photographs; direct measurement of stone study models and digital subtraction of 3D models, showing that the most reliable method to measure the differences in VD was the digital subtraction of 3D models. This method could detect whether the occlusion returned to its pre-crown state regarding the overbite and also gave an indication of appropriate follow-up timeframe to evaluate this resolution.

These are preliminary results and the pilot study was designed to guide future research. There were no previous reliable data regarding the evaluation of VD and its effects when this pilot study was conducted. A random sample size was selected to give insight to build a future power calculation for future studies. The investigators would like to continue this pilot work and carry out a full study recruiting children that are assigned to receive a HTPMC during routine appointments in the DDS.

By understanding where occlusal compensation occurs in the mouth following placement of a HTPMC, and how long this takes to occur, more accurate information can be given to parents on what to expect following treatment, supporting joint treatment planning and decision making regarding the dental care of the child. In addition, where more than one crown is required, treatment planning can be timed more precisely to ensure future treatment is carried out at the optimal time.

DETAILED DESCRIPTION:
This is a prospective observational cohort study involving children undergoing treatment at Dundee Dental Hospital & School. The study involves taking additional measurements of children who have already had treatment planned that includes a HTPMC (having a crown placed over a decayed tooth).

There will be no interventions or invasive procedures as part of this study. As an additional procedure, specific to this study (not included in the standard care), participants will have dental impressions taken to compare pre and post HTPMC placement (right after the treatment and at 2, 4, 6, and 8 weeks follow-up) state of their mouths. Dental impressions are a routine procedure that children regularly undergo for orthodontic treatment or to make mouth guards for sports.

Children having a HTPMC fitted would not have a dental impression taken before and after the HTPMC placement or at subsequent appointments as part of standard care.

Since the aim is to track the changes that happen in children's mouth, the investigators are going to use these extra procedures of taking dental impressions to analyse digitally (by making a 3D scan of the stone study models). This will allow us to see how long it takes for the children's vertical dimension to come back to its pre-treatment state and what the changes are that happen in their mouth after the placement of a HTPMC.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 5 to 9 years old
* children who are eligible to receive a HTPMC to manage primary molars carious lesions;
* children who have not had a HTPMC fitted within the last 6 weeks;
* children who understand what is involved in the study and have signed and given assent to participate;
* children that can cooperate with dental care including having a dental impression taken; and
* children whose parents are willing and able to attend the follow-up appointments 2, 4, 6 and 8 weeks after the treatment.

Exclusion Criteria:

* children who do not have parental agreement to participate; or
* children who have self-reported occlusal parafunctional habits (e.g. bruxism, constantly open mouths).

Individuals will not be enrolled to the study if they are participating in the clinical phase of another interventional trial/study or have done so within the last 30 days. Individuals who are participating in the follow-up phase of another interventional trial/study, or who are enrolled in an observational study, will be co-enrolled where the Chief Investigators of each study agree that it is appropriate.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from 5 to 9 years old undergoing dental treatments at Children's Clinic in Dundee Dental Hospital & School, University of Dundee
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
The height of the crowned tooth and its opposing tooth. | Immediately after, at 2, 4, 6 and 8 weeks following placement of the Hall Technique Preformed Metal Crown.
  Changes in teeth height will be measured in millimetres using a digital software.

SECONDARY OUTCOMES:
Height difference in the crowned tooth and the vertical dimension. | Immediately after, at 2, 4, 6 and 8 weeks following placement of the Hall Technique Preformed Metal Crown.
  Measured by the increase in the height of canines on stone study models in millimetres using a digital software.
The difference in height of the crowned tooth, the opposing and adjacent teeth. | Immediately after, at 2, 4, 6 and 8 weeks following placement of the Hall Technique Preformed Metal Crown.
  Teeth height will be measured in millimetres using a digital software.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Araujo, Principal Investigator — University of Dundee/University of São Paulo
Locations (1):
- University of Dundee, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludwig KH, Fontana M, Vinson LA, Platt JA, Dean JA. The success of stainless steel crowns placed with the Hall technique: a retrospective study. J Am Dent Assoc. 2014 Dec;145(12):1248-53. doi: 10.14219/jada.2014.89. PMID 25429038
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] So D, Evans DJ, Borrie F, Roughley M, Lamont T, Keightley A, Innes NPT: Measurement of occlusal equilibration following Hall crown placement - a pilot study (abstract). J Dent Res 2015;94(spec. issue A):0080.
- [Result] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395